CLINICAL TRIAL: NCT00037427
Title: Airway Responses Following Chlorine Gas Exposure
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 1170; R01HL069664 (NIH)
Record Dates: First submitted 2002-05-16; First posted 2002-05-17 (Estimated); Last update posted 2016-03-16 (Estimated); Status verified 2005-05

CONDITIONS: Asthma; Lung Diseases
MeSH Terms: conditions — Asthma; Lung Diseases

SUMMARY:
To determine lung airway responses following chlorine gas exposure.

DETAILED DESCRIPTION:
DESIGN NARRATIVE:

The specific aims of the study are to determine: (1) the effects of asthma with pre-existing airway hyper reactivity on the pulmonary function and airway reactivity and inflammation responses to chlorine; (2) the effects of chlorine concentration on the pulmonary function and airway reactivity and inflammation responses to chlorine; and (3) to assess the time dynamics of the pulmonary function and airway reactivity and inflammation responses to chlorine. It is hypothesized that both airway hyperactivity and higher chlorine concentration will result in larger changes in pulmonary function and airway reactivity and inflammation responses, and that these changes will have differential time courses following chlorine exposure. This study uses two controlled human exposure experiments, utilizing a single-blind, repeated-measures, and counter- balanced design. The two subject groups for both experiments will consist of 21 individuals with no airway hyperactivity, and 21 individuals with both asthma and airway hyperactivity. In Experiment One, subjects are exposed for 15 minutes separately to each of: (1) chlorine at 0.4 ppm; (2) chlorine at 1.0 ppm; and (3) filtered air (Control). Pulmonary function and airway reactivity are measured immediately pre-exposure and 1 and 20 hours post-exposure. Airway inflammation, as determined by cellular and biochemical components from sputum-induction, is measured 65 hours pre-exposure and 20 hours post-exposure. In Experiments Two, subjects are exposed for 15 minutes separately to each of: (1) chlorine (concentration determined from Experiment One); (2) filtered air (Control). Pulmonary function and airway reactivity are measured immediately pre-exposure and at 3 and 72 hours post-exposure. Sputum-induction is performed 65 hours pre-exposure and at 3 and 72 hours post-exposure. The results of this study will provide information on a major irritant chemical relevant to occupational environments. Specially, the susceptibility of a large sub-population at increased risk, the dose-response effects, and the post-exposure time dynamics of the effects of chlorine gas will be determined.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2001-09; Study Completion 2004-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Colin Solomon — University of California at San Francisco